CLINICAL TRIAL: NCT02041468
Title: A Phase IV Multicenter Trial to Evaluate the Resistance Mechanisms and Real-world Pharmacoeconomics of Crizotinib and Its Companion Diagnostic Test in Advanced ALK-positive Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: Study to Evaluate Resistance Mechanisms and Real-world Pharmacoeconomics of Crizotinib in NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: Pfizer (Industry); Quebec Clinical Research Organization in Cancer (Other); PeriPharm (Other); Personalized Medicine Partnership for Cancer (Other)
Responsible Party: Principal Investigator, Dr. Jason Agulnik, Principal Investigator, Jewish General Hospital
Other Study IDs: Q-CROC-05
Record Dates: First submitted 2013-12-20; First posted 2014-01-22 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: ALK-positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will collect plasma, platelet-depleted plasma, tumor tissue (biopsy of a metastatic site that has acquired resistant to treatment) and primary archived tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pharmacoeconomic main study: Patients from Quebec and Ontario (first or second line treatment)
- Biomarker sub-study: Patients from Quebec only (first or second line treatment)

SUMMARY:
This is a phase IV multicenter trial to evaluate the mechanisms of resistance and pharmacoeconomic (PE) impact of crizotinib and its companion diagnostic test used in a real-life setting in advanced ALK-positive non-small cell lung cancer (NSCLC) patients.

The study will address two anticipated issues surrounding personalized medicine and treatment with crizotinib:

* it will enable real-life Heath Economics and Outcome Research (HEOR)
* it will validate and/or identify new blood-based or tissue-based biomarkers of resistance to crizotinib.

At least 30 patients will be recruited in Quebec and Ontario for the PE study. Patients will be asked to complete quality-of-life questionnaires at regular intervals in a real-life setting of treatment with crizotinib.

Approximately 25 patients will be recruited to the biomarker sub-study in Quebec to understand resistance mechanisms of crizotinib. In these patients, a biopsy from any accessible metastatic lesion will be obtained when the patient is no longer responding to treatment, as well as blood sampling during regular treatment visits.

DETAILED DESCRIPTION:
This is a phase IV multicenter trial to evaluate the mechanisms of resistance and pharmacoeconomic (PE) impact of crizotinib and its companion diagnostic test used in a real-life setting in advanced ALK-positive non-small cell lung cancer (NSCLC) patients.

NSCLC represent 80% of all new cases of lung cancer. One molecular subtype of NSCLC is the ALK-positive subtype. The anaplastic lymphoma kinase (ALK) is a transmembrane receptor tyrosine kinase. Activation of ALK occurs through the formation of gene fusions and in NSCLC, the gene fusion partner for ALK is primarily EML4. The resulting fusion protein is capable of activating the ALK kinase domain, leading to cell growth. The estimated prevalence for ALK rearrangements in NSCLC is 3-5%, and is more commonly found amongst patients with adenocarcinoma histology, in never smokers and in those who are known to be wild type for EGFR and KRAS.

Crizotinib is a potent inhibitor of ALK and is approved for the treatment of advanced ALK+ NSCLC patients. This is an example of personalized medicine, where patients are selected for treatment based upon a molecular assay, and are provided a specific therapy (crizotinib) for their disease. The pharmacoeconomic impact of using genetic information in early treatment decisions in NSCLC has not been determined. Despite the benefits of crizotinib, some patients do not respond to treatment and most patients will eventually develop resistance. To date, it is unclear why some rare patients do not respond to treatment and the resistance mechanisms of crizotinib have not been fully elucidated.

The study will address two anticipated issues surrounding personalized medicine and treatment with crizotinib:

* it will enable real-life Heath Economics and Outcome Research (HEOR)
* it will validate and/or identify new blood-based or tissue-based biomarkers of resistance to crizotinib.

At least 30 patients will be recruited in Quebec and Ontario for the PE study. Patients will be asked to complete quality-of-life questionnaires at regular intervals in a real-life setting of treatment with crizotinib.

Approximately 25 patients will be recruited to the biomarker sub-study in Quebec to understand resistance mechanisms of crizotinib. In these patients, a biopsy from any accessible metastatic lesion will be obtained when the patient is no longer responding to treatment, as well as blood sampling during regular treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed locally advanced or metastatic NSCLC
* Presence of the ALK-fusion oncogene (ALK+) as determined using a validated testing platform
* Measurable disease according to RECIST v. 1.1
* Planned or ongoing treatment with crizotinib
* Signed and dated IRB-approved informed consent document
* Ability to read and understand English or French
* 18 years of age or older

Exclusion Criteria:

* Acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease.
* Unwilling to provide consent for genetic studies of the tumor, whole blood, or plasma specimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) found positive for ALK mutation from participating hospitals in Quebec.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The pharmacoeconomic impact of using personalized medicine for the treatment of ALK+ lung cancer. | From the date of registration until date of death from any cause, assessed up to 60 months.
  Pharmacoeconomic impact (cost-effectiveness and cost utility) will be evaluated by questionnaires completed by the patient and caregiver. These include quality of life, health resource utilization, work productivity and activity impairment, and health questionnaires

SECONDARY OUTCOMES:
Type of resistance mechanisms identified in crizotinib-resistant tumors | At progression of disease, an expected average of 24 months.
  A biopsy will be taken from a metastatic lesion that has progressed despite treatment with crizotinib. Genomic material will be isolated and sequenced to identify causes of acquired resistance to crizotinib.
Change in blood-based biomarkers of response to crizotinib. | From the date of registration until the date of treatment discontinuation, an expected average of 24 months.
  Plasma will be isolated from patients pre-treatment, at every disease assessment, at progression of disease, and at treatment discontinuation. This will be used to identify changes in blood-based biomarkers using proteomics analysis by mass spectrometry.
Number of participants with adverse events related to the biopsy procedure. | Up to 4 years.
  Adverse events possibly, probably or definitely related to the biopsy procedure will be reported according to the The NCI's Common Toxicity Criteria version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jason Agulnik, MD, Principal Investigator — Jewish General Hospital; Victor Cohen, MD, Principal Investigator — Jewish General Hospital
Locations (8):
- Canada (8):
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center (JGH, St-Mary's, MGH, RVH), Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - CSSS Rimouski, Rimouski, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Institut Universitaire de cardiologie et de pneumonologie, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Katayama R, Shaw AT, Khan TM, Mino-Kenudson M, Solomon BJ, Halmos B, Jessop NA, Wain JC, Yeo AT, Benes C, Drew L, Saeh JC, Crosby K, Sequist LV, Iafrate AJ, Engelman JA. Mechanisms of acquired crizotinib resistance in ALK-rearranged lung Cancers. Sci Transl Med. 2012 Feb 8;4(120):120ra17. doi: 10.1126/scitranslmed.3003316. Epub 2012 Jan 25. PMID 22277784
- [Background] Camidge DR, Doebele RC. Treating ALK-positive lung cancer--early successes and future challenges. Nat Rev Clin Oncol. 2012 Apr 3;9(5):268-77. doi: 10.1038/nrclinonc.2012.43. PMID 22473102
- [Background] Kwak EL, Bang YJ, Camidge DR, Shaw AT, Solomon B, Maki RG, Ou SH, Dezube BJ, Janne PA, Costa DB, Varella-Garcia M, Kim WH, Lynch TJ, Fidias P, Stubbs H, Engelman JA, Sequist LV, Tan W, Gandhi L, Mino-Kenudson M, Wei GC, Shreeve SM, Ratain MJ, Settleman J, Christensen JG, Haber DA, Wilner K, Salgia R, Shapiro GI, Clark JW, Iafrate AJ. Anaplastic lymphoma kinase inhibition in non-small-cell lung cancer. N Engl J Med. 2010 Oct 28;363(18):1693-703. doi: 10.1056/NEJMoa1006448. PMID 20979469
- [Background] Doebele RC, Pilling AB, Aisner DL, Kutateladze TG, Le AT, Weickhardt AJ, Kondo KL, Linderman DJ, Heasley LE, Franklin WA, Varella-Garcia M, Camidge DR. Mechanisms of resistance to crizotinib in patients with ALK gene rearranged non-small cell lung cancer. Clin Cancer Res. 2012 Mar 1;18(5):1472-82. doi: 10.1158/1078-0432.CCR-11-2906. Epub 2012 Jan 10. PMID 22235099
- [Derived] Couetoux du Tertre M, Marques M, McNamara S, Gambaro K, Hoffert C, Tremblay L, Bouchard N, Diaconescu R, Blais N, Couture C, Pelsser V, Wang H, McIntosh L, Hindie V, Parent S, Cortes L, Breton YA, Pottiez G, Croteau P, Higenell V, Izzi L, Spatz A, Cohen V, Batist G, Agulnik J. Discovery of a putative blood-based protein signature associated with response to ALK tyrosine kinase inhibition. Clin Proteomics. 2020 Feb 7;17:5. doi: 10.1186/s12014-020-9269-6. eCollection 2020. PMID 32055239